CLINICAL TRIAL: NCT01330329
Title: Comparison of a Traditional Behavioral Weight Loss Program Versus a Technology - Based Weight Loss Program in Severely Obese Individuals
Brief Title: Comparison of Weight Loss Programs for Individuals With Severe Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Jessica Unick, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0209-10
Record Dates: First submitted 2011-04-05; First posted 2011-04-06 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight loss; Exercise; Intervention studies
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Serum Bactericidal Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBT + technology system (SBT+FIT) (Experimental): Participants will receive a standard behavioral weight loss program and will also be asked to use the Body Media FIT system as part of their weight loss intervention.
  Interventions: Behavioral: SBT + technology system (SBT+FIT)
- Standard behavioral treatment (SBT) (Experimental): Participants receive a standard behavioral weight loss program similar to that used in other large trials such as Look AHEAD and the Diabetes Prevention Program.
  Interventions: Behavioral: Standard behavioral treatment

INTERVENTIONS:
Behavioral: Standard behavioral treatment — Participants receive a standard behavioral weight loss program similar to that used in other large trials such as Look AHEAD and the Diabetes Prevention Program. Individuals will come to weekly group meetings for 6-months and will be instructed to reduce caloric intake, increase physical activity, and self-monitor their weight, eating, and exercise behaviors.
  Arms: Standard behavioral treatment (SBT)
Behavioral: SBT + technology system (SBT+FIT) — Participants will receive a standard behavioral weight loss program and will also be asked to use the Body Media FIT system as part of their weight loss intervention. Individuals will come to weekly group meetings for 6-months and will be instructed to reduce caloric intake, increase physical activity, and self-monitor their weight, eating, and exercise behaviors. Participants in this group will also wear an armband that measures energy expenditure and they will log their food intake on the internet.
  Arms: SBT + technology system (SBT+FIT)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a technology-based system (the Body Media FIT system) for enhancing weight loss in severely obese individuals (BMI: ≥ 40 kg/m2). The investigators will compare two 6-month interventions: 1) a standard behavioral weight loss program (SBT) and 2) a standard behavioral weight loss program plus the use of the Body Media FIT system (SBT+FIT). The Body Media® FIT system is a novel weight loss tool consisting of an armband that measures energy expenditure, a digital display watch that provides "real time" physical activity and energy expenditure feedback, and access to a system website which allows individuals to track their food intake and set exercise and dietary goals. We will examine differences in physical activity, weight loss, and program adherence between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-55
* Body mass index (BMI) ≥40kg/m2 (or no more than 440 lbs)

Exclusion Criteria:

* Recent weight loss (≥ 10 pounds within the past 6 months)
* Currently pregnant, pregnant within the last 6 months, or planning on becoming pregnant in the next 6 months.
* Presence of any condition that would limit exercise participation (assessed by the Physical Activity Readiness Questionnaire (PAR-Q)).
* A history of myocardial infarction or other heart-related surgeries.
* Currently enrolled in a commercial weight loss program.
* A recent (< 1 year) diagnosis or hospitalization for a psychological condition or history of psychosis (e.g. - Schizophrenia, Bipolar, Eating Disorder)
* Diagnosed with cancer within the past year or currently undergoing cancer treatment.
* Currently taking weight loss medications.
* Currently do not have daily access to a computer or Internet.
* Individuals with diabetes

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 6-months

SECONDARY OUTCOMES:
Change in physical activity | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Rena Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Unick JL, O'Leary KC, Dorfman L, Thomas JG, Strohacker K, Wing RR. Consistency in compensatory eating responses following acute exercise in inactive, overweight and obese women. Br J Nutr. 2015 Apr 14;113(7):1170-7. doi: 10.1017/S000711451500046X. Epub 2015 Mar 17. PMID 25778833